CLINICAL TRIAL: NCT01964495
Title: Reduction of Antibiotic Therapy by Biomakers in Patients With CAP Episodes (REDUCE Study)
Acronym: REDUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Collaborators: Foreest Medical School (Unknown); Pulmoscience (Unknown)
Responsible Party: Principal Investigator, W.G.Boersma, MSc, MD, PhD, Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Duijkers
Record Dates: First submitted 2013-09-30; First posted 2013-10-17 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Common clinical practice (Active Comparator): Treatment according to current guidelines. Often a 7 day course of antibiotics. Initial treatment should be broad spectrum antibiotics and can be narrowed down if a specific pathogen is identified.
  Interventions: Drug: Treatment according to current guidelines
- CRP-guided treatment (Experimental): Treatment according to CRP levels. Patients will be started on broad spectrum antibiotics for at least 3 days, treatment can be switched to small-spectrum antibiotics if a specific pathogen is identified. From day 4 to 7 daily blood tests will be performed in order to evaluate whether or not treatment can be discontinued. If treatment is discontinued, no more blood tests will be performed.
  Interventions: Drug: Discontinuation of treatment according to CRP levels
- PCT guided treatment (Experimental): Treatment according to PCT levels. Patients will be started on broad spectrum antibiotics for at least 3 days, treatment can be switched to small-spectrum antibiotics if a specific pathogen is identified. From day 4 to 7 daily blood tests will be performed in order to evaluate whether or not treatment can be discontinued. If treatment is discontinued, no more blood tests will be performed.
  Interventions: Drug: Discontinuation of treatment according to PCT levels

INTERVENTIONS:
Drug: Discontinuation of treatment according to CRP levels — The cutoff point is a CRP below 100 mg/L and a reduction to 50% of the initial value.
  Other Names: Broad spectrum antibiotics; Small spectrum antibiotics
  Arms: CRP-guided treatment
Drug: Discontinuation of treatment according to PCT levels — The cutoff point is a PCT below 0.25 mcg/L or a reduction to 10% of the initial value.
  Other Names: Broad spectrum antibiotics; Small spectrum antibiotics
  Arms: PCT guided treatment
Drug: Treatment according to current guidelines — Often a 7 days course of antibiotics, treatment may be extended if the attending physician deems it necessary.
  Other Names: Broad spectrum antibiotics; Small spectrum antibiotics
  Arms: Common clinical practice

SUMMARY:
The purpose of this study is to evaluate two different treatment strategies in patients admitted to hospital with Community Acquired Pneumonia. The investigators hypothesize treatment according to both procalcitonin (PCT) and C-reactive protein (CRP) will be effective in reducing the length of antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients with a diagnosis of CAP and all criteria listed below:

1. Age 18 or above, no upper age limit will be employed.
2. Patients must require hospitalisation.
3. Clinical presentation of an acute illness with one or more of the following symptoms:

   1. Temperature ≥ 38.0 ⁰C (100.4°F)
   2. Dyspnoea
   3. Cough (with or without expectoration of sputum)
   4. Chest pain
   5. Malaise or fatigue
   6. Myalgia
   7. Gastro-intestinal symptoms
   8. Rales, rhonchi or wheezing
   9. Egophony or bronchial breath sounds
4. New consolidation(s) on the chest radiograph.
5. Written informed consent obtained.
6. (Pre-event) Life expectancy > 30 days

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. (Severe) immunosuppression (e.g. HIV infection, chemotherapy, use of immunosuppressants).
2. Active neoplastic disease.
3. Obstruction pneumonia (e.g. from lung cancer).
4. Aspiration pneumonia.
5. Pneumonia that developed within 8 days after hospital discharge.
6. Unable and/or unlikely to comprehend and/or follow the protocol.
7. Pregnant and/or lactating women.
8. Other infection that requires treatment with antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Length of antibiotic treatment | End of the study

SECONDARY OUTCOMES:
Length of stay | End of the study
Clinical response | End of the study
  Cure - resolution or improvement of symptoms and clinical signs related to pneumonia without the need for additional or alternative antibiotic therapy
  Failure - persistence or progression of all signs and symptoms of the acute process after randomisation or the development of a new pulmonary or extrapulmonary respiratory tract infection, or the progression of abnormalities on chest radiograph after randomisation, or death due to pneumonia, or the inability to complete the study owing to adverse events
  Indeterminate - patient receives less than 80% of the study drug for reasons other than clinical failure, a concomitant infection outside the respiratory tract requiring antibiotic treatment, lost to follow-up, or death unrelated to the primary diagnosis.
30-day mortality | End of the study, periodically by the DSMB
  All cause
Time to clinical stability | End of the study
  Patients are considered clinically stable if they fulfill all of these criteria: Temperature equal to or below 37.8 degrees celsius, heart rate equal to or below 100 beats per minute, respiratory rate equal to or below 24 breaths per minute, systolic blood pressure equal to or above 90 mmHg, arterial oxygen saturation equal to or above 90 percent or pO2 equal to or above 60 mmHg on room air, ability to maintain oral intake, normal mental status.
Relapse rate | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ruud Duijkers, MSc, MD, Study Director — Medisch Centrum Alkmaar; Wim G Boersma, MD, PhD, MSc, Principal Investigator — Medisch Centrum Alkmaar; Dominic Snijders, MSc, PhD, MD, Study Chair — Slotervaart ziekenhuis
Locations (3):
- Netherlands (3):
  - Medical Centre Alkmaar, Alkmaar, North Holland
  - Slotervaart Hospital, Amsterdam, North Holland
  - ISALA clinics, Zwolle, Overijssel

REFERENCES:
- [Derived] Hessels L, Duijkers R, Schoorl M, Terpstra L, Thijs W, Boersma W. The Value of Soluble Urokinase Plasminogen Activator Receptor (suPAR) as Predictive Tool in Hospitalised Patients With Community-Acquired Pneumonia (CAP). Clin Respir J. 2025 Jun;19(6):e70089. doi: 10.1111/crj.70089. PMID 40523722
- [Derived] Duijkers R, Prins HJ, Kross M, Snijders D, van den Berg JWK, Werkman GM, van der Veen N, Schoorl M, Bonten MJM, van Werkhoven CH, Boersma WG. Biomarker guided antibiotic stewardship in community acquired pneumonia: A randomized controlled trial. PLoS One. 2024 Aug 20;19(8):e0307193. doi: 10.1371/journal.pone.0307193. eCollection 2024. PMID 39163362